CLINICAL TRIAL: NCT00002284
Title: A Pilot Study To Evaluate Azidothymidine (AZT) in the Treatment of Human Immunodeficiency Virus (HIV) Infection in Patients Receiving a Bone Marrow Transplant
Brief Title: A Study of Azidothymidine (AZT) in the Treatment of HIV Infection in Patients Receiving a Bone Marrow Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014A; 006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: Lymphoma, Large-Cell; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Bone Marrow Transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Dendritic Cell Sarcoma, Interdigitating; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine whether zidovudine (AZT) in conjunction with bone marrow transplantation prevents the reinfection of donor hematopoietic/lymphoid cells in patients with positive HTLV III antibody and large cell/diffuse histiocytic lymphoma. Patients who are candidates will be evaluated for HTLV III activity and drug levels.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with current life-threatening infection at time of transplant that would preclude a transplant are excluded.

Concurrent Medication:

Excluded:

* Other anti-retroviral agents.

Patients with current life-threatening infection at time of transplant that would preclude a transplant are excluded.

Patients must be:

* HTLV III antibody positive by ELISA or Western blot or HTLV III viremia.
* At high mortal risk with a diagnosis of AIDS or AIDS Related Complex (ARC).
* Also patient must fall into one of the following categories:
* Have an HIV seronegative identical twin to serve as a bone marrow donor.
* Have documentation of large cell/diffuse histiocytic lymphoma/DPDL.
* Be a good risk candidate for bone marrow transplant.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hemapheresis Treatment Ctr, Baltimore, Maryland, United States